CLINICAL TRIAL: NCT01303445
Title: Drug-drug Interaction Study of the Effect of Omeprazole 80 mg q.d. at Steady State on the Pharmacokinetics and Pharmacodynamics of Aggrenox® Every 12 Hours at Steady State in Healthy Male and Female Volunteers (an Open-label, Randomised, Crossover Study)
Brief Title: Drug-drug Interaction Study of Aggrenox and Omeprazole in Normal Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 9.197
Record Dates: First submitted 2011-02-23; First posted 2011-02-24 (Estimated); Results first posted 2012-07-24 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2012-07

CONDITIONS: Healthy
MeSH Terms: interventions — Aspirin, Dipyridamole Drug Combination; Omeprazole

ARMS (4):
- Treatment A (Active Comparator): Aggrenox alone
  Interventions: Drug: Aggrenox alone
- Treatment B (Experimental): Aggrenox and omeprazole
  Interventions: Drug: Aggrenox and omeprazole
- Treatment C (Active Comparator): Omeprazole alone
  Interventions: Drug: Omeprazole alone
- Treatment D (Experimental): Aggrenox and omeprazole
  Interventions: Drug: Aggrenox and omeprazole

INTERVENTIONS:
Drug: Aggrenox alone — Aggrenox 1 capsule twice daily for 7 days
  Arms: Treatment A
Drug: Aggrenox and omeprazole — Aggrenox 1 capsule twice daily and omeprazole 80mg once daily for 7 days
  Arms: Treatment B
Drug: Aggrenox and omeprazole — Aggrenox 1 capsule twice daily and omeprazole 80mg once daily for 7 days
  Arms: Treatment D
Drug: Omeprazole alone — omeprazole 80 once daily for 7 days
  Arms: Treatment C

SUMMARY:
The objective of the current study is to investigate if a drug-drug interaction occurs with the administration of omeprazole 80 mg q.d. at steady state on the pharmacokinetics of dipyridamole and the pharmacodynamics of ASA-induced platelet aggregation inhibition (components of Aggrenox®) when administered every 12 hours at steady state.

DETAILED DESCRIPTION:
Purpose:

ELIGIBILITY:
Inclusion criteria:

1. Healthy males and females according to the following criteria:

   Based upon a complete medical history, including the physical examination, vital signs (blood pressure(BP), pulse rate (PR)), 12-lead ECG, clinical laboratory tests
2. BMI >18.5 and BMI <32 kg/m2 (Body Mass Index)

Exclusion criteria:

1. Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance in the opinion of the PI
2. Any evidence of a clinically relevant concomitant disease
3. Clinically significant gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological, hormonal, or hematologic (including a history of abnormal bruising) disorders in the opinion of the PI
4. Surgery of the gastrointestinal tract that might impair drug absorption
5. Clinically significant diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
6. History of relevant orthostatic hypotension, fainting spells or blackouts.
7. Chronic or relevant acute infections
8. History of relevant allergy/hypersensitivity (including allergy to study drugs or its excipients, or reactions to related drugs [e.g., non-steroidal anti-inflammatory drugs])
9. Intake of drugs with a long half-life (¿24 hours) within one month, or less than 10 half lives of the respective drug, prior to study drug administration or during the trial
10. Use of drugs which might reasonably influence the results of the trial (including OTC antacids) based on the knowledge at the time of protocol preparation within 14 days prior to administration or during the trial
11. Participation in another trial with an investigational drug within two months prior to administration or during the trial
12. Tobacco use within the 90 days prior to check-in and throughout the study
13. Alcohol abuse within the past 2 years
14. Drug abuse within the past 2 years
15. Blood donation or other significant blood loss within 56 days (inclusive) prior to screening, or plasma donation within 7 days (inclusive) prior to study drug administration, or during the trial
16. Excessive physical activities (within one week prior to first drug administration or during the trial)
17. Any laboratory value outside the reference range that is of clinical relevance in the opinion of the PI; including positive virology, or urine drug screen, or positive fecal occult blood test
18. Inability to comply with dietary regimen of trial site
19. In the opinion of the investigator it would be in the best interest of the subject to be excluded from participation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2011-03; Primary Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 9.197.001 Boehringer Ingelheim Investigational Site, Tempe, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- ABCD Sequence: Aggrenox/Aggrenox+Omeprazole/Omeprazole/Aggrenox+Omeprazole
- CDAB Sequence: Omeprazole/Aggrenox+Omeprazole/Aggrenox/Aggrenox+Omeprazole
Period: First Intervention (7 Days)
Arm/Group | ABCD Sequence | CDAB Sequence
Started | 30 | 30
Completed | 29 | 30
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Second Intervention (7 Days)
Arm/Group | ABCD Sequence | CDAB Sequence
Started | 29 | 30
Completed | 28 | 28
Not Completed | 1 | 2
Not completed — Adverse Event | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0
Period: Washout (14 Days)
Arm/Group | ABCD Sequence | CDAB Sequence
Started | 28 | 28
Completed | 27 | 26
Not Completed | 1 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 0 | 2
Period: Third Intervention (7 Days)
Arm/Group | ABCD Sequence | CDAB Sequence
Started | 27 | 26
Completed | 27 | 26
Not Completed | 0 | 0
Period: Fourth Intervention (7 Days)
Arm/Group | ABCD Sequence | CDAB Sequence
Started | 27 | 26
Completed | 26 | 26
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Follow-up Period (14 Days)
Arm/Group | ABCD Sequence | CDAB Sequence
Started | 26 | 26
Completed | 26 | 25
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Arm/Group | Entire Study Population
Number analyzed (Participants) | 60
Age, Continuous [Mean (Full Range); unit: years] | 35.3 [20 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 48
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 57
  Black / African American | 3
Weight [Mean (Full Range); unit: kilograms] | 75.69 [55.2 to 101.7]
Body Mass Index (BMI) [Mean (Full Range); unit: kilograms per square meter] | 26.81 [20.45 to 31.94]

OUTCOME MEASURES:

1. Primary Outcome: Plasma Dipyridamole Maximum Concentration (Cmax)
Description: Maximum measured concentration of dipyridamole in plasma
Time Frame: 7 days
Population: The pharmacokinetic data set (PK set) and the pharmacodynamic data set (PD set) include all treated subjects with data that do not have a relevant protocol violation (relevant to PK or PD). No data collected for Omeprazole arm since no plasma dipyridamole was expected for this treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter
Groups:
- Aggrenox Alone BID: Aggrenox (aspirin/extended release dipyridamole) 25mg/200mg capsules BID (twice daily)
- Aggrenox BID Plus Omeprazole QD Following Aggrenox Alone: Aggrenox 25mg/200mg capsules BID plus Omeprazole 40mg QD (once daily) following Aggrenox alone
- Aggrenox BID Plus Omeprazole QD Following Omeprazole Alone: Aggrenox 25mg/200mg capsules BID plus Omeprazole 40mg QD (once daily) following Omeprazole alone
- Omeprazole Alone QD: Omeprazole 40mg QD (once daily)
Arm/Group | Aggrenox Alone BID | Aggrenox BID Plus Omeprazole QD Following Aggrenox Alone | Aggrenox BID Plus Omeprazole QD Following Omeprazole Alone | Omeprazole Alone QD
Number analyzed (Participants) | 55 | 54 | 54 | 0
nanogram/milliliter | 2750 (30.4) | 2550 (27.5) | 2550 (29.1) |
Statistical Analysis 1: Comparison: Aggrenox Alone BID vs Aggrenox BID Plus Omeprazole QD Following Omeprazole Alone; Comparison of Aggrenox + Omeprazole following Omeprazole versus Aggrenox alone; Test type: Non-Inferiority or Equivalence — Bioequivalence was established if the 90% confidence interval of the mean ratio fell within the 80 to 125% target range; Percent Mean Ratio = 92.03, 90% CI [86.95 to 97.40]
Statistical Analysis 2: Comparison: Aggrenox Alone BID vs Aggrenox BID Plus Omeprazole QD Following Aggrenox Alone; Comparison of Aggrenox + Omeprazole following Aggrenox versus Aggrenox alone; Test type: Non-Inferiority or Equivalence — Bioequivalence was established if the 90% confidence interval of the mean ratio fell within the 80 to 125% target range; Percent Mean Ratio = 92.30, 90% CI [87.76 to 97.08]

2. Primary Outcome: Plasma Dipyridamole Area Under Plasma Concentration-time Curve From Zero to 12 Hours (AUC0-12)
Description: Area under the concentration time curve of the analyte in plasma from 0 to 12 hours at steady state
Time Frame: 7 days
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (nanogram/milliliter)*hours
Arm/Group | Aggrenox Alone BID | Aggrenox BID Plus Omeprazole QD Following Aggrenox Alone | Aggrenox BID Plus Omeprazole QD Following Omeprazole Alone | Omeprazole Alone QD
Number analyzed (Participants) | 55 | 53 | 54 | 0
(nanogram/milliliter)*hours | 17100 (33.7) | 16700 (28.4) | 16500 (31.1) |
Statistical Analysis 1: Comparison: Aggrenox Alone BID vs Aggrenox BID Plus Omeprazole QD Following Omeprazole Alone; Comparison of Aggrenox + Omeprazole following Omeprazole versus Aggrenox alone; Test type: Non-Inferiority or Equivalence — Bioequivalence was established if the 90% confidence interval of the mean ratio fell within the 80 to 125% target range; Percent Mean Ratio = 96.38, 90% CI [90.96 to 102.13]
Statistical Analysis 2: Comparison: Aggrenox Alone BID vs Aggrenox BID Plus Omeprazole QD Following Aggrenox Alone; Comparison of Aggrenox + Omeprazole following Aggrenox versus Aggrenox alone; Test type: Non-Inferiority or Equivalence — Bioequivalence was established if the 90% confidence interval of the mean ratio fell within the 80 to 125% target range; Percent Mean Ratio = 97.03, 95% CI [93.26 to 100.95]

3. Primary Outcome: Inhibition of Platelet Aggregation at 4 Hours Post Dose (IPA4)
Description: IPA4 equals the platelet aggregation measured 4 hours post dose divided by the platelet aggregation measured at baseline (multiplied by 100).
Time Frame: 7 days
Population: The pharmacokinetic data set (PK set) and the pharmacodynamic data set (PD set) include all treated subjects with data that do not have a relevant protocol violation (relevant to PK or PD). No data collected for Omeprazole arm since no platelet inhibition was expected for this treatment.
Measure: Mean (Standard Deviation); unit: percent of baseline platelet aggregation
Arm/Group | Aggrenox Alone BID | Aggrenox BID Plus Omeprazole QD Following Aggrenox Alone | Aggrenox BID Plus Omeprazole QD Following Omeprazole Alone | Omeprazole Alone QD
Number analyzed (Participants) | 55 | 54 | 54 | 0
percent of baseline platelet aggregation | 97.89 (2.74) | 96.34 (4.21) | 97.02 (2.69) |
Statistical Analysis 1: Comparison: Aggrenox Alone BID vs Aggrenox BID Plus Omeprazole QD Following Omeprazole Alone; Comparison of Aggrenox + Omeprazole following Omeprazole versus Aggrenox alone; Test type: Non-Inferiority or Equivalence — Bioequivalence was established if the 90% confidence interval of the mean ratio fell within the 80 to 125% target range; Percent Mean Ratio = 99.02, 90% CI [98.32 to 99.72]
Statistical Analysis 2: Comparison: Aggrenox Alone BID vs Aggrenox BID Plus Omeprazole QD Following Aggrenox Alone; Comparison of Aggrenox + Omeprazole following Aggrenox versus Aggrenox alone; Test type: Non-Inferiority or Equivalence — Bioequivalence was established if the 90% confidence interval of the mean ratio fell within the 80 to 125% target range; Percent Mean Ratio = 98.42, 90% CI [97.66 to 99.18]

4. Secondary Outcome: Plasma Dipyridamole Minimum Concentration (Cmin)
Description: Minimum measured concentration of dipyridamole in plasma
Time Frame: 7 days
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter
Arm/Group | Aggrenox Alone BID | Aggrenox BID Plus Omeprazole QD Following Aggrenox Alone | Aggrenox BID Plus Omeprazole QD Following Omeprazole Alone | Omeprazole Alone QD
Number analyzed (Participants) | 55 | 54 | 54 | 0
nanogram/milliliter | 679 (47.1) | 723 (41.8) | 713 (46.5) |
Statistical Analysis 1: Comparison: Aggrenox Alone BID vs Aggrenox BID Plus Omeprazole QD Following Omeprazole Alone; Comparison of Aggrenox + Omeprazole following Omeprazole versus Aggrenox alone; Test type: Non-Inferiority or Equivalence — Bioequivalence was established if the 90% confidence interval of the mean ratio fell within the 80 to 125% target range; Percent Mean Ratio = 105.55, 90% CI [97.09 to 114.74]
Statistical Analysis 2: Comparison: Aggrenox Alone BID vs Aggrenox BID Plus Omeprazole QD Following Aggrenox Alone; Comparison of Aggrenox + Omeprazole following Aggrenox versus Aggrenox alone; Test type: Non-Inferiority or Equivalence — Bioequivalence was established if the 90% confidence interval of the mean ratio fell within the 80 to 125% target range; Percent Mean Ratio = 106.09, 90% CI [98.64 to 114.09]

5. Secondary Outcome: Inhibition of Platelet Aggregation at 12 Hours Post Dose (IPA12)
Description: IPA12 equals the platelet aggregation measured 12 hours post dose divided by the platelet aggregation measured at baseline (multiplied by 100).
Time Frame: 7 days
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent of baseline platelet aggregation
Arm/Group | Aggrenox Alone BID | Aggrenox BID Plus Omeprazole QD Following Aggrenox Alone | Aggrenox BID Plus Omeprazole QD Following Omeprazole Alone | Omeprazole Alone QD
Number analyzed (Participants) | 55 | 54 | 54 | 0
percent of baseline platelet aggregation | 98.78 (2.53) | 97.80 (3.00) | 98.11 (2.98) |
Statistical Analysis 1: Comparison: Aggrenox Alone BID vs Aggrenox BID Plus Omeprazole QD Following Omeprazole Alone; Comparison of Aggrenox + Omeprazole following Omeprazole versus Aggrenox alone; Test type: Non-Inferiority or Equivalence — Bioequivalence was established if the 90% confidence interval of the mean ratio fell within the 80 to 125% target range; Percent Mean Ratio = 99.38, 90% CI [98.80 to 99.95]
Statistical Analysis 2: Comparison: Aggrenox Alone BID vs Aggrenox BID Plus Omeprazole QD Following Aggrenox Alone; Comparison of Aggrenox + Omeprazole following Aggrenox versus Aggrenox alone; Test type: Non-Inferiority or Equivalence — Bioequivalence was established if the 90% confidence interval of the mean ratio fell within the 80 to 125% target range; Percent Mean Ratio = 99.02, 90% CI [98.46 to 99.59]

6. Secondary Outcome: Percentage Peak-to-trough Fluctuation (%PTF)
Description: PTF = 100*((Cmax-Cmin)/Cavg) where Cavg=(AUC0-12)/12.
Time Frame: 7 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent of average hourly plasma conc.
Arm/Group | Aggrenox Alone BID | Aggrenox BID Plus Omeprazole QD Following Aggrenox Alone | Aggrenox BID Plus Omeprazole QD Following Omeprazole Alone | Omeprazole Alone QD
Number analyzed (Participants) | 55 | 53 | 54 | 0
percent of average hourly plasma conc. | 144 (31.8) | 132 (41.4) | 134 (41.2) |

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Aggrenox Alone BID | Aggrenox BID Plus Omeprazole QD Following Aggrenox Alone | Omeprazole Alone QD | Aggrenox BID Plus Omeprazole QD Following Omeprazole Alone
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/55 | 0/57 | 0/57
Other Adverse Events (participants affected / at risk) | 41/56 | 15/55 | 17/57 | 48/57
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aggrenox Alone BID (N=56) | Aggrenox BID Plus Omeprazole QD Following Aggrenox Alone (N=55) | Omeprazole Alone QD (N=57) | Aggrenox BID Plus Omeprazole QD Following Omeprazole Alone (N=57)
Palpitations (Cardiac disorders) | 3 | 0 | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 3 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 4 | 2 | 6
Flatulence (Gastrointestinal disorders) | 0 | 1 | 3 | 0
Nausea (Gastrointestinal disorders) | 19 | 0 | 4 | 14
Vomiting (Gastrointestinal disorders) | 12 | 2 | 2 | 14
Chest discomfort (General disorders) | 6 | 1 | 1 | 4
Chills (General disorders) | 1 | 1 | 3 | 1
Contusion (Injury, poisoning and procedural complications) | 3 | 2 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 4 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 18 | 4 | 2 | 20
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 2 | 1
Dizziness (Nervous system disorders) | 7 | 3 | 2 | 10
Headache (Nervous system disorders) | 39 | 6 | 7 | 41
Paraesthesia (Nervous system disorders) | 3 | 0 | 2 | 1
Somnolence (Nervous system disorders) | 1 | 1 | 4 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 | 1 | 0 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other - Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.